CLINICAL TRIAL: NCT03726034
Title: Life Story Work for Promoting Relationship Between Older Adults and live-in Migrant Caregivers: a Randomized Controlled Feasibility Trail
Brief Title: Life Story Book for Older Adults and live-in Migrant Caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tung Wah College (Other)
Responsible Party: Principal Investigator, Ken HM HO, Assistant Professor, Tung Wah College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RESC2018013
Record Dates: First submitted 2018-10-22; First posted 2018-10-31 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Home Caregiver-older Adults Relationship
Keywords: Caregiver relationship; Life story book; migrant caregivers; older adults; randomized controlled trial

STUDY DESIGN:
Intervention Model Description: Two-arm single-blinded randomized controlled feasibility trial.
Who Masked: Outcomes Assessor
Masking Description: A trained research assistant will be responsible to collect demographic data and assessing the outcomes at T0, T1, T2. The research assistant will be blinded to the grouping of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Life story book training (Experimental): The migrant caregivers will receive training (six weekly 1.5-hour sessions) about life story approach by a part-time trained interventionist with psychology or social work background with at least three years of working experience working with older people and have basic knowledge about the life story work. After training, the migrant caregivers will be asked to produce the life story book individually at home with the older adults
  Interventions: Behavioral: Life Story Book
- Communication skills training (Active Comparator): The migrant caregivers who have randomly assigned into the control group will receive communication skills training (two 1.5-hour sessions) offered by another trained interventionist with psychology or social work background with at least three years of working experience working with older people. They would not receive any additional training on life story work.
  Interventions: Behavioral: Self-selected social activities

INTERVENTIONS:
Behavioral: Life Story Book — The protocol of life story book creation is validated in Hong Kong. The life story book would contain two elements: (1) the development of the older adults over the course of his/her lifetime (i.e. from childhood to old age); and (2) the psychosocial development and ways of life of the older adults (e.g. education, marriage, career, and hobbies). The product of the intervention will be a written story with pictures or other memorabilia that are meaningful to the older adults. There is no limitation on the number of words, pages, and pictures. Four to six 60-minute scheduled sessions will be needed for the older adult and the live-in migrant caregivers to discuss and produce the lifestory book at home.
  Arms: Life story book training
Behavioral: Self-selected social activities — To control the possible social interaction effects on the dyadic relationship and wellbeing, the caregivers of the control group will conduct self-selected social activities with older adult at home individually for four times weekly.
  Arms: Communication skills training

SUMMARY:
The relationship between older adults and live-in migrant caregivers is always challenged by weak emotional connectedness, ineffective communication, power struggling and unmet needs of both, that may lead to poor care quality and negatively influence their well-being. The aim of this study is to explore the feasibility to train live-in migrant caregivers to adopt Life Story Work for promoting the dyadic relationship with the older adults, through communication and negotiation, mutual understanding and expression of needs. This is a two-arm randomized controlled trial. The caregivers of the intervention group will receive training on life story work. Then they will be asked to create a life storybook of the older adult at home individually, with the support from the team. The caregivers in the control group will receive training on communication skills only, and will be asked to conduct social activities at home. Outcomes such as quality of relationship; well-being, depressive symptoms and level of loneliness of the older adults; and job satisfaction of the caregivers will be assessed at baseline, post-intervention and 3 months follow up. Focus group interviews will be conducted with the caregivers of the intervention group for soliciting their comments regarding to the intervention.

DETAILED DESCRIPTION:
There are approximately 21.5 million live-in migrant workers, and around 41% of them are employed in Asia. Among the 352 thousand live-in migrant workers in Hong Kong, at least 21% of them are caregivers of older adults. The 2016 Policy Address suggested a pilot scheme for training live-in migrant caregivers to take care of the older people in Hong Kong to meet the trend of Ageing in Place, and cope with the dreadful shortage of formal long-term care services. As such, Social Welfare Department of Hong Kong is now implementing an 18-month pilot scheme to train live-in migrant workers to care for older adults in order to improve the well-being of the older adults. However, there is no effective evidence-based intervention available for such caregiving arrangement, not only locally but also internationally. The common training for live-in migrant workers is about instrumental training, such as feeding and bathing. According to the Relationship-Centred Care Model, relationship is the core for good quality of care. Life story work have been tested effective in various settings for promoting the psychological well-being of older adults with/out dementia, as well as proven useful in promoting mutual understanding and communication between caregivers and care-recipients.

The project is of value in that:

* It is a pioneer study, which aims to promote relationship between live-in migrant caregivers and older adults to support good quality of care.
* The life story work is a skill that is easily learnt and adopted for promoting and sustaining good relationship that may impact on the well-being of caregivers and care-recipients.
* Reduce the needs of formal long-term care services by retaining the older adults to be cared at home.
* The life story work has a potential to be adopted by all types of caregivers (including formal and informal caregivers; live-in and live-out) for promoting the caregiver-care recipient dyadic relationship through communication and negotiation between the dyads, mutual understanding and expression of needs.

Objectives:

1. Explore the feasibility to train live-in migrant caregivers to adopt life story work;
2. Explore the feasibility of trained live-in migrant caregivers to produce a life story book with the older adult at home; and
3. Provide preliminary evidence of efficacy of the life story work on improving dyadic relationship, psychosocial outcomes of the older adults, and satisfaction of caregivers.

ELIGIBILITY:
Older adults:

Inclusion Criteria:

* aged 60 or above
* community dwelling
* being cared by participating migrant caregivers

Exclusion Criteria:

* unwilling to create life story book with the migrant caregivers
* not verbally communicable
* diagnosed with serious psychiatric illnesses or terminal illnesses

Migrant caregivers:

Inclusion Criteria:

* have been working for the older adutls for more than 6 months
* at least completed primary education
* be communicable in either English or Cantonese.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The change in quality of migrant caregiver-older adults relationship as assessed by 4-item Lawrence quality of the caregiver-care recipient relationship scale | basline (T0), immediately post-intervention (T1), 3-month follow up (T2)
  General closeness, communication, similarity of views about life, and degree of getting along will be captured. Total score of the scale ranges from 4-16. Higher values represent a better quality of relationship. The cronhach's alpha for this scale was 0.85.

SECONDARY OUTCOMES:
The change in loneliness of the older adults as assessed by the Chinese version of 6-item De Jong Gierveld Loneliness Scale | basline (T0), immediately post-intervention (T1), 3-month follow up (T2)
  The scale consists of two sub-scales: emotional and social loneliness. Cronbach's alpha for this scale was 0.76. The overall loneliness score ranges from 0 to 6, where 0 means no loneliness and 6 indicates severe loneliness.
The change in depressive symptoms of the older adults as assessed by the Chinese version of 15-item Geriatric Depression Scale | basline (T0), immediately post-intervention (T1), 3-month follow up (T2)
  The 15 items are scored on a dichotomous scale, from 0 to 1. Total score of the scale ranges from 0-15. Higher values represent the older adult has more depressive symptoms. A cutoff of greater or equals to 8 identifies clinically significant depression in older adults.
The change in well-being of the dyad as assessed by the 12-item General Health Questionnaire | basline (T0), immediately post-intervention (T1), 3-month follow up (T2)
  Total score of he scale ranges from 0-36. Higher values represent the participant has worse health. The coefficient alpha for this scale was 0.87.
The change in satisfaction of caregiver as assessed by the 6-item Care Work Satisfaction Scale | basline (T0), immediately post-intervention (T1), 3-month follow up (T2)
  The 6 items are rated on a ordinal scale from strongly disagree to strongly agree.

OTHER OUTCOMES:
The change in dependency level of older adult as assessed by the 11-item Modified Barthel Index | basline (T0), immediately post-intervention (T1), 3-month follow up (T2)
  The total score of the index ranges from 0-105. Higher values represent the older adult is more independent. The coefficient alpha was 0.92.

IPD SHARING:
Plan to Share IPD: No
The data to be shared will include the measured outcomes.

REFERENCES:
- [Background] Lai CKY, Igarashi A, Yu CTK, Chin KCW. Does life story work improve psychosocial well-being for older adults in the community? A quasi-experimental study. BMC Geriatr. 2018 May 16;18(1):119. doi: 10.1186/s12877-018-0797-0. PMID 29769035

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT03726034/Prot_SAP_000.pdf